CLINICAL TRIAL: NCT05181189
Title: NMDA Enhancement Combined With Omega-3 Fatty Acids for the Treatment of Early Dementia
Brief Title: NMDA Enhancement Combined With Omega-3 for Early Dementia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-0510163
Record Dates: First submitted 2021-12-23; First posted 2022-01-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Omega 3 Fatty Acids; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAOIB+Omega-3 (Experimental)
  Interventions: Drug: DAOIB+Omega-3
- DAOIB+Placebo (Placebo Comparator)
  Interventions: Drug: DAOIB+Placebo

INTERVENTIONS:
Drug: DAOIB+Omega-3 — The omega-3 fatty acids dose will be adjusted every 8 weeks according to clinical evaluation.
  Arms: DAOIB+Omega-3
Drug: DAOIB+Placebo — Placebo
  Arms: DAOIB+Placebo

SUMMARY:
In this 4-year proposed project, we will enroll 140 patients with aMCI or mild AD into a 24-week randomized, double-blind, placebo-controlled drug trial. All patients will be allocated randomly to one of two treatment groups for 24 weeks (n = 70 in each group) in a double-blind manner: [1] DAOIB + omega-3; [2] DAOIB + placebo. We will assess the patients every 8 weeks during the treatment period (weeks 0, 8, 16, and 24). We hypothesize that DAOIB combined with omega-3 will yield better efficacy than placebo in improving the cognitive function, global functioning and quality of life in patients with aMCI or mild AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease or mild cognitive impairment
* MMSE between 10-26
* CDR 1 or 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* memantine or special omega-3 fatty acids therapy within 3 months before enrollment
* Severe visual or hearing impairment

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Alzheimer's disease assessment scale-cognitive subscale scores range from 0 (best) to 70 (worst)

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24 | week 8, 16, 24
  Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24
Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24 | week 0, 8, 16, 24
  Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24
Change from baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) at week 8, 16 and 24 | week 0, 8, 16, 24
  Change from baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) at week 8, 16 and 24
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 8, 16 and 24 | week 0, 8, 16, 24
  The assessment appears to be a suitable instrument for evaluating activities of daily living in early-phase dementia. Its scores range from 0 (worst) to 78 (best)
Change from baseline in Quality of life score at week 8, 16 and 24 | week 0, 8, 16, 24
  Quality of life will be assessed by Medical Outcomes Study Short-Form-36 (SF-36). The SF-36 consists of eight sections: (1) vitality, (2) physical functioning, (3) bodily pain, (4) general health perceptions, (5) physical role functioning, (6) emotional role functioning, (7) social role functioning, and (8) mental health.
Change from baseline in the composite score of a battery of additional cognitive tests at week 24 | week 0, 24
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (Wechsler Memory Scale, Spatial Span), verbal/nonverbal learning and memory tests (Wechsler Memory Scale, Word Listing).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No